CLINICAL TRIAL: NCT04199117
Title: Centralized Health System Interventions to Enhance Reach: A Factorial Screening Experiment
Brief Title: Health Systems Reach Interventions Project
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2019-0939; 2P01CA180945-06 (NIH); A534253 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*G (Other: UW Madison); 5736 (Other: NIH 2P01CA180945-06 Sub-Project ID); UW20070 (Other: UW Madison); Protocol Version 10/25/2023 (Other: UW Madison)
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-01

CONDITIONS: Smoking, Cigarette; Smoking Cessation
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Intervention Model Description: 2 x 2 x 2 x 2 factorial experiment
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors collecting follow-up data on quit attempts, use of treatment, and smoking status will be blind to experimental condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (16):
- Incentive,Tailored,Care Manage,Intensive Treatment (Experimental): Participants randomly assigned to this condition will have access to incentives for completing a first smoking cessation counseling call up to 4 times over 2 years, will receive 5 tailored letters promoting use of smoking cessation treatment over 2 years, will receive 5 Tobacco Care Management support and motivational encouragement calls over 2 years, and will have access to 3 smoking cessation quit counseling calls and 12-weeks of either combination nicotine replacement or varenicline up to 4 times over 2 years.
  Interventions: Drug: Varenicline; Drug: Combination nicotine patch and nicotine mini-lozenge treatment; Behavioral: Monetary incentives for initiating treatment; Behavioral: Automated tailored outreach; Behavioral: Care management; Behavioral: Multiple smoking cessation coaching calls
- Incentive,Tailored,Care Manage,Standard Treatment (Experimental): Participants randomly assigned to this condition will have access to incentives for completing a first smoking cessation counseling call up to 4 times over 2 years, will receive 5 tailored letters promoting use of smoking cessation treatment over 2 years, will receive 5 Tobacco Care Management support and motivational encouragement calls over 2 years, and will have access to standard smoking cessation treatment (referral to the state tobacco quitline and/or their primary care provider) over 2 years.
  Interventions: Behavioral: Monetary incentives for initiating treatment; Behavioral: Automated tailored outreach; Behavioral: Care management; Other: Wisconsin Tobacco Quit Line referral; Other: Primary care provider referral
- Incentive,Tailored,No Care Manage,Intensive Treatment (Experimental): Participants randomly assigned to this condition will have access to incentives for completing a first smoking cessation counseling call up to 4 times over 2 years, will receive 5 tailored letters promoting use of smoking cessation treatment over 2 years, will not receive Tobacco Care Management support and motivational encouragement calls, and will have access to 3 smoking cessation quit counseling calls and 12-weeks of either combination nicotine replacement or varenicline up to 4 times over 2 years.
  Interventions: Drug: Varenicline; Drug: Combination nicotine patch and nicotine mini-lozenge treatment; Behavioral: Monetary incentives for initiating treatment; Behavioral: Automated tailored outreach; Behavioral: Multiple smoking cessation coaching calls
- Incentive,Tailored,No Care Manage,Standard Treatment (Experimental): Participants randomly assigned to this condition will have access to incentives for completing a first smoking cessation counseling call up to 4 times over 2 years, will receive 5 tailored letters promoting use of smoking cessation treatment over 2 years, will not receive Tobacco Care Management support and motivational encouragement calls, and will have access to standard smoking cessation treatment (referral to the state tobacco quitline and/or their primary care provider) over 2 years.
  Interventions: Behavioral: Monetary incentives for initiating treatment; Behavioral: Automated tailored outreach; Other: Wisconsin Tobacco Quit Line referral; Other: Primary care provider referral
- Incentive,Untailored,Care Manage,Intensive Treatment (Experimental): Participants randomly assigned to this condition will have access to incentives for completing a first smoking cessation counseling call up to 4 times over 2 years, will receive 5 untailored letters promoting use of smoking cessation treatment over 2 years, will receive 5 Tobacco Care Management support and motivational encouragement calls over 2 years, and will have access to 3 smoking cessation quit counseling calls and 12-weeks of either combination nicotine replacement or varenicline up to 4 times over 2 years.
  Interventions: Drug: Varenicline; Drug: Combination nicotine patch and nicotine mini-lozenge treatment; Behavioral: Monetary incentives for initiating treatment; Behavioral: Care management; Behavioral: Untailored outreach; Behavioral: Multiple smoking cessation coaching calls
- Incentive,Untailored,Care Manage,Standard Treatment (Experimental): Participants randomly assigned to this condition will have access to incentives for completing a first smoking cessation counseling call up to 4 times over 2 years, will receive 5 untailored letters promoting use of smoking cessation treatment over 2 years, will receive 5 Tobacco Care Management support and motivational encouragement calls over 2 years, and will have access to standard smoking cessation treatment (referral to the state tobacco quitline and/or their primary care provider) over 2 years.
  Interventions: Behavioral: Monetary incentives for initiating treatment; Behavioral: Care management; Other: Wisconsin Tobacco Quit Line referral; Other: Primary care provider referral; Behavioral: Untailored outreach
- Incentive,Untailored,No Care Manage,Intensive Treatment (Experimental): Participants randomly assigned to this condition will have access to incentives for completing a first smoking cessation counseling call up to 4 times over 2 years, will receive 5 untailored letters promoting use of smoking cessation treatment over 2 years, will not receive Tobacco Care Management support and motivational encouragement calls, and will have access to 3 smoking cessation quit counseling calls and 12-weeks of either combination nicotine replacement or varenicline up to 4 times over 2 years.
  Interventions: Drug: Varenicline; Drug: Combination nicotine patch and nicotine mini-lozenge treatment; Behavioral: Monetary incentives for initiating treatment; Behavioral: Untailored outreach; Behavioral: Multiple smoking cessation coaching calls
- Incentive,Untailored,No Care Manage,Standard Treatment (Experimental): Participants randomly assigned to this condition will have access to incentives for completing a first smoking cessation counseling call up to 4 times over 2 years, will receive 5 untailored letters promoting use of smoking cessation treatment over 2 years, will not receive Tobacco Care Management support and motivational encouragement calls, and will have access to standard smoking cessation treatment (referral to the state tobacco quitline and/or their primary care provider) over 2 years.
  Interventions: Behavioral: Monetary incentives for initiating treatment; Other: Wisconsin Tobacco Quit Line referral; Other: Primary care provider referral; Behavioral: Untailored outreach
- No Incentive,Tailored,Care Manage,Intensive Treatment (Experimental): Participants randomly assigned to this condition will have not access to incentives for completing smoking cessation counseling, will receive 5 tailored letters promoting use of smoking cessation treatment over 2 years, will receive 5 Tobacco Care Management support and motivational encouragement calls over 2 years, and will have access to 3 smoking cessation quit counseling calls and 12-weeks of either combination nicotine replacement or varenicline up to 4 times over 2 years.
  Interventions: Drug: Varenicline; Drug: Combination nicotine patch and nicotine mini-lozenge treatment; Behavioral: Automated tailored outreach; Behavioral: Care management; Behavioral: Multiple smoking cessation coaching calls
- No Incentive,Tailored,Care Manage,Standard Treatment (Experimental): Participants randomly assigned to this condition will not have access to incentives for completing smoking cessation counseling, will receive 5 tailored letters promoting use of smoking cessation treatment over 2 years, will receive 5 Tobacco Care Management support and motivational encouragement calls over 2 years, and will have access to standard smoking cessation treatment (referral to the state tobacco quitline and/or their primary care provider) over 2 years.
  Interventions: Behavioral: Automated tailored outreach; Behavioral: Care management; Other: Wisconsin Tobacco Quit Line referral; Other: Primary care provider referral
- No Incentive,Tailored,No Care Manage,Intensive Treatment (Experimental): Participants randomly assigned to this condition will not have access to incentives for completing smoking cessation counseling, will receive 5 tailored letters promoting use of smoking cessation treatment over 2 years, will not receive Tobacco Care Management support and motivational encouragement calls, and will have access to 3 smoking cessation quit counseling calls and 12-weeks of either combination nicotine replacement or varenicline up to 4 times over 2 years.
  Interventions: Drug: Varenicline; Drug: Combination nicotine patch and nicotine mini-lozenge treatment; Behavioral: Automated tailored outreach; Behavioral: Multiple smoking cessation coaching calls
- No Incentive,Tailored,No Care Manage,Standard Treatment (Experimental): Participants randomly assigned to this condition will not have access to incentives for completing smoking cessation counseling, will receive 5 tailored letters promoting use of smoking cessation treatment over 2 years, will not receive Tobacco Care Management support and motivational encouragement calls, and will have access to standard smoking cessation treatment (referral to the state tobacco quitline and/or their primary care provider) over 2 years.
  Interventions: Behavioral: Automated tailored outreach; Other: Wisconsin Tobacco Quit Line referral; Other: Primary care provider referral
- No Incentive,Untailored,Care Manage,Intensive Treatment (Experimental): Participants randomly assigned to this condition will not have access to incentives for completing smoking cessation counseling, will receive 5 untailored letters promoting use of smoking cessation treatment over 2 years, will receive 5 Tobacco Care Management support and motivational encouragement calls over 2 years, and will have access to 3 smoking cessation quit counseling calls and 12-weeks of either combination nicotine replacement or varenicline up to 4 times over 2 years.
  Interventions: Drug: Varenicline; Drug: Combination nicotine patch and nicotine mini-lozenge treatment; Behavioral: Care management; Behavioral: Untailored outreach; Behavioral: Multiple smoking cessation coaching calls
- No Incentive,Untailored,Care Manage,Standard Treatment (Experimental): Participants randomly assigned to this condition will not have access to incentives for completing smoking cessation counseling, will receive 5 untailored letters promoting use of smoking cessation treatment over 2 years, will receive 5 Tobacco Care Management support and motivational encouragement calls over 2 years, and will have access to standard smoking cessation treatment (referral to the state tobacco quitline and/or their primary care provider) over 2 years.
  Interventions: Behavioral: Care management; Other: Wisconsin Tobacco Quit Line referral; Other: Primary care provider referral; Behavioral: Untailored outreach
- No Incentive,Untailored,No Care Manage,IntensiveTreatment (Experimental): Participants randomly assigned to this condition will not have access to incentives for completing smoking cessation counseling, will receive 5 untailored letters promoting use of smoking cessation treatment over 2 years, will not Tobacco Care Management support and motivational encouragement calls, and will have access to 3 smoking cessation quit counseling calls and 12-weeks of either combination nicotine replacement or varenicline up to 4 times over 2 years.
  Interventions: Drug: Varenicline; Drug: Combination nicotine patch and nicotine mini-lozenge treatment; Behavioral: Untailored outreach; Behavioral: Multiple smoking cessation coaching calls
- No Incentive,Untailored,No Care Manage,Standard Treatment (Active Comparator): Participants randomly assigned to this condition will not have access to incentives for completing smoking cessation counseling, will receive 5 untailored letters promoting use of smoking cessation treatment over 2 years, will not receive Tobacco Care Management support and motivational encouragement calls, and will have access to standard smoking cessation treatment (referral to the state tobacco quitline and/or their primary care provider) over 2 years.
  Interventions: Other: Wisconsin Tobacco Quit Line referral; Other: Primary care provider referral; Behavioral: Untailored outreach

INTERVENTIONS:
Drug: Varenicline — Participants randomized to intensive treatment who choose to use this intervention will receive one 0.5 mg pill for the first 3 days, starting 7 days prior to the target quit day (TQD). They will then use one 0.5 mg pill twice daily for the next 4 days. After the first week of study medication ramp up, participants will use one 1 mg pill twice daily until 11 weeks post-TQD. This will not be used at the same time as combination nicotine replacement therapy.
  Arms: Incentive,Tailored,Care Manage,Intensive Treatment; Incentive,Tailored,No Care Manage,Intensive Treatment; Incentive,Untailored,Care Manage,Intensive Treatment; Incentive,Untailored,No Care Manage,Intensive Treatment; No Incentive,Tailored,Care Manage,Intensive Treatment; No Incentive,Tailored,No Care Manage,Intensive Treatment; No Incentive,Untailored,Care Manage,Intensive Treatment; No Incentive,Untailored,No Care Manage,IntensiveTreatment
Drug: Combination nicotine patch and nicotine mini-lozenge treatment — Participants randomized to intensive treatment who choose to use this intervention will receive 12 weeks of nicotine patches and nicotine mini-lozenges starting on the target quit day (TQD). Participants who smoke more than 10 cigarettes/day will start with a 21 mg patch for 8 weeks, and then titrate down to a 14 mg patch for 2 weeks and then a 7 mg patch for 2 weeks. Participants who smoke 5-10 cigarettes/day will be given 10 weeks of 14 mg patches and then 2 weeks of 7 mg patches. Participants will receive 2 mg mini-lozenges for use starting on the target quit date and the following 12 weeks. Participants will be instructed to use 9-20 mini-lozenges per day (one every 1-2 hours) for the first 6 weeks, then reduce to a mini-lozenge every 2-4 hours for 3 weeks, and then a mini-lozenge every 4-8 hours for 3 weeks. Combination nicotine patch and nicotine mini-lozenge treatment will not be used at the same time as varenicline.
  Arms: Incentive,Tailored,Care Manage,Intensive Treatment; Incentive,Tailored,No Care Manage,Intensive Treatment; Incentive,Untailored,Care Manage,Intensive Treatment; Incentive,Untailored,No Care Manage,Intensive Treatment; No Incentive,Tailored,Care Manage,Intensive Treatment; No Incentive,Tailored,No Care Manage,Intensive Treatment; No Incentive,Untailored,Care Manage,Intensive Treatment; No Incentive,Untailored,No Care Manage,IntensiveTreatment
Behavioral: Monetary incentives for initiating treatment — Participants randomized to this intervention will earn an incentive each time they complete a first counseling session in an available treatment, up to 2 rounds of counseling per year, and up to 4 rounds of counseling over 2 years of enrollment.
  Arms: Incentive,Tailored,Care Manage,Intensive Treatment; Incentive,Tailored,Care Manage,Standard Treatment; Incentive,Tailored,No Care Manage,Intensive Treatment; Incentive,Tailored,No Care Manage,Standard Treatment; Incentive,Untailored,Care Manage,Intensive Treatment; Incentive,Untailored,Care Manage,Standard Treatment; Incentive,Untailored,No Care Manage,Intensive Treatment; Incentive,Untailored,No Care Manage,Standard Treatment
Behavioral: Automated tailored outreach — Participants randomized to this intervention will receive 5 tailored letters delivered every 4-6 months. Letter content will be tailored to participant demographics and use of study treatment, and personalized with references to their primary care teams and tobacco care manager. Letters offer encouragement to quit and information about how to access available treatments.
  Arms: Incentive,Tailored,Care Manage,Intensive Treatment; Incentive,Tailored,Care Manage,Standard Treatment; Incentive,Tailored,No Care Manage,Intensive Treatment; Incentive,Tailored,No Care Manage,Standard Treatment; No Incentive,Tailored,Care Manage,Intensive Treatment; No Incentive,Tailored,Care Manage,Standard Treatment; No Incentive,Tailored,No Care Manage,Intensive Treatment; No Incentive,Tailored,No Care Manage,Standard Treatment
Behavioral: Care management — Participants randomized to this intervention will receive 5 live, proactive phone calls lasting 10-15 minutes from as assigned Tobacco Care Manager who will provide manualized support and motivational encouragement, discuss available treatment options, and inform the participant how to initiate treatment when ready to quit.
  Arms: Incentive,Tailored,Care Manage,Intensive Treatment; Incentive,Tailored,Care Manage,Standard Treatment; Incentive,Untailored,Care Manage,Intensive Treatment; Incentive,Untailored,Care Manage,Standard Treatment; No Incentive,Tailored,Care Manage,Intensive Treatment; No Incentive,Tailored,Care Manage,Standard Treatment; No Incentive,Untailored,Care Manage,Intensive Treatment; No Incentive,Untailored,Care Manage,Standard Treatment
Other: Wisconsin Tobacco Quit Line referral — This is recommended standard care that will be offered to participants who are not medically eligible for varenicline or combination nicotine patch or who are randomized to standard treatment access. The Wisconsin Tobacco Quit Line (WTQL) offers a single 20-minute counseling session to all Wisconsin residents ready to set a date to stop smoking in the next month, at no charge, and offers those who meet their medical eligibility criteria a 2-week supply of either nicotine patches, lozenges, or gums, at no charge. The WTQL assumes full clinical responsibility for participants' use of cessation medications dispensed by the WTQL.
  Arms: Incentive,Tailored,Care Manage,Standard Treatment; Incentive,Tailored,No Care Manage,Standard Treatment; Incentive,Untailored,Care Manage,Standard Treatment; Incentive,Untailored,No Care Manage,Standard Treatment; No Incentive,Tailored,Care Manage,Standard Treatment; No Incentive,Tailored,No Care Manage,Standard Treatment; No Incentive,Untailored,Care Manage,Standard Treatment; No Incentive,Untailored,No Care Manage,Standard Treatment
Other: Primary care provider referral — This is a form of recommended standard care that will be offered to participants who are not medically eligible for varenicline or combination nicotine patch or who are randomized to standard treatment access. Participants who choose to use this intervention will be referred electronically to their primary care provider for counseling and/or medication if they express an interest in quitting in the next 30 days and agree to this referral.
  Arms: Incentive,Tailored,Care Manage,Standard Treatment; Incentive,Tailored,No Care Manage,Standard Treatment; Incentive,Untailored,Care Manage,Standard Treatment; Incentive,Untailored,No Care Manage,Standard Treatment; No Incentive,Tailored,Care Manage,Standard Treatment; No Incentive,Tailored,No Care Manage,Standard Treatment; No Incentive,Untailored,Care Manage,Standard Treatment; No Incentive,Untailored,No Care Manage,Standard Treatment
Behavioral: Untailored outreach — Participants randomized to this intervention will receive 5 untailored letters delivered every 4-6 months. Letter content will not be tailored or personalized. Letters will offer information about how to access available treatments.
  Arms: Incentive,Untailored,Care Manage,Intensive Treatment; Incentive,Untailored,Care Manage,Standard Treatment; Incentive,Untailored,No Care Manage,Intensive Treatment; Incentive,Untailored,No Care Manage,Standard Treatment; No Incentive,Untailored,Care Manage,Intensive Treatment; No Incentive,Untailored,Care Manage,Standard Treatment; No Incentive,Untailored,No Care Manage,IntensiveTreatment; No Incentive,Untailored,No Care Manage,Standard Treatment
Behavioral: Multiple smoking cessation coaching calls — Participants randomized to intensive treatment access who choose to quit will receive three 15-20-minute quit coaching calls from a trained smoking cessation health counselor. Calls will be scheduled for one week pre-quit, one day after the target quit day, and one week after the target quit day.
  Arms: Incentive,Tailored,Care Manage,Intensive Treatment; Incentive,Tailored,No Care Manage,Intensive Treatment; Incentive,Untailored,Care Manage,Intensive Treatment; Incentive,Untailored,No Care Manage,Intensive Treatment; No Incentive,Tailored,Care Manage,Intensive Treatment; No Incentive,Tailored,No Care Manage,Intensive Treatment; No Incentive,Untailored,Care Manage,Intensive Treatment; No Incentive,Untailored,No Care Manage,IntensiveTreatment

SUMMARY:
This project seeks to identify ways to enhance the reach of evidence-based smoking cessation treatments among adult primary care patients who smoke daily and are not ready to start treatment at study enrollment. The 2x2x2x2 factorial experiment will evaluate the extent to which 4 intervention components promote the use of evidence-based treatments to help smokers not initially ready to quit to cease smoking over 2 years. The intervention components tested include: modest financial incentives for completing an initial counseling session in a smoking cessation treatment (vs. none); automated semi-annual outreach materials sent via patients' preferred communication modality using data in the electronic health record to tailor and personalize invitations to use available treatments to quit smoking (vs. untailored letters); direct, proactive telephone outreach from a tobacco care manager who will promote treatment use and deliver motivational intervention twice per year (vs. none); and access to 3 no-cost telephone smoking cessation counseling calls with combination nicotine replacement therapy (C-NRT) or varenicline (vs. state tobacco quitline and primary care provider referral). Proactive treatment offers will be made up to 22 months after enrollment. Smoking status and use of any smoking cessation treatments will be assessed every 6 months through 2 years of study enrollment. Data from 1664 adult primary care patients meeting inclusion/exclusion criteria will be analyzed to see whether the intervention components have an effect on the use of treatment (primary outcome) and smoking status after 2 years of treatment access (secondary outcome). The project will evaluate the manipulated intervention components first in terms of treatment initiation (defined as rates of completing at least 1 smoking cessation counseling session prior to a target stop-smoking date), and then in terms of end-of-study (2 year post-enrollment) abstinence rates (secondary outcome), and cost-effectiveness in promoting reach (tertiary outcome). This experiment will help to identify health system reach interventions that effectively enhance utilization of stop smoking treatments in an effort to help more smokers quit and to prevent tobacco-induced cancer morbidity and mortality.

DETAILED DESCRIPTION:
Design and Objective: This 2-year experimental study will evaluate the effectiveness, costs, and cost-effectiveness of four interventions designed to connect primary care patients who smoke with evidence-based stop-smoking treatment. The interventions to be tested are healthcare system interventions intended to better attract patients who smoke to stop-smoking treatments that work. Participants enrolled in the study will be randomized to 1 level of each of the following 4 intervention components: 1) to receive financial incentive each time they complete a first counseling telephone call in a new round of stop-smoking treatment (for up to 4 rounds of treatment) or no incentives for starting treatment; 2) to receive tailored letters encouraging use of evidence-based stop-smoking treatment every 4-6 months for 2 years, or non-tailored letters every 4-6 months for 2 years; 3) to receive calls every 4-6 months from a Tobacco Care Manager who will provide motivational counseling to patients to encourage them to use stop-smoking treatment, and will connect patients willing to quit with available treatments, or no Tobacco Care Manager calls; and 4) access to intensive treatment (standard 12-week regimens of 2 nicotine medications used together, also called combination nicotine replacement therapy, or varenicline, a non-nicotine pill), with 3 telephone counseling sessions, all of which improve stop-smoking success rates), or standard care (referral to a quitline offering telephone counseling and 2 weeks of one nicotine medication provided by the quitline, and referral to the patient's primary care provider). The objective is to identify the intervention components and combination of components that best promote use of smoking cessation treatment and tobacco abstinence.

Recruitment and Participants: Participants will be 1664 primary care patients recruited through their primary care clinics in 2 healthcare systems in central and eastern Wisconsin. At the launch of recruitment in a clinic, all patients known to smoke at that clinic will receive notice that a new tobacco specialist, a Tobacco Care Manager, is available to help them quit smoking and given information about how to contact them. At healthcare visits, patients will be asked if they smoke, and if they do, told that the clinic has a new program for smokers that will start with a phone call from a Tobacco Care Manager within the next few days. Patients will be able to opt out of receiving such calls if they do not want them. The Tobacco Care Manager will offer information to all patients who smoke about resources available to help them quit smoking, and will ask them if they are interested in a research study. For those not willing to quit within a month and interested in the study, the Tobacco Care Manager will describe this study and ask them if they want to be screened for eligibility for the study. Those who assent to and pass the screening will then be given detailed information about the study and asked to provide informed consent for participation. For those who consent to participation, the Tobacco Care Manager will administer a 10-15-minute baseline interview over the phone, randomize patients to experimental condition, and inform them of the types of stop-smoking information and resources they will receive over the course of the 2-year study. Everyone in the study will receive a letter about their randomly assigned smoking cessation resources and study information by mail after enrollment and 4 more times over the next 2 years. Follow-up assessments will occur every 6 months over 2 years to see if participants are still smoking, if they have tried to quit, and if they have used any stop-smoking treatment. One and two years after enrollment, some participants will be asked to come to their clinic for breath and urine tests to determine if they are still smoking. Patients may be asked to complete additional follow-up calls if they start stop-smoking treatment, to see if they are smoking, using treatment, experiencing withdrawal, and are still motivated and confident about quitting and treatment at 3, 12, and 26 weeks after trying to quit smoking.

Outcomes and Analyses. The primary outcome of interest in this study is whether or not participants use the stop-smoking treatments available to them. The primary research question of interest is the extent to which each intervention improves the reach of stop-smoking treatments (i.e., how many people use the treatment), and whether particular packages of interventions do this particularly well. A second important research question is whether the study interventions help more people stop smoking during the 2-year study, and which packages of interventions do this well. A third question of importance to healthcare systems that may adopt these interventions is whether the interventions are affordable and whether or not they improve treatment use rates and tobacco abstinence rates in a manner that is cost-effective. Total costs of each intervention component will be estimated and used to compute costs per reach (initiating treatment), per quit (achieving abstinence), and per quality-adjusted life-year gained, and to estimate the net monetary benefit and incremental cost effectiveness ratio for each intervention component and combination of components.

Knowledge to be Gained. This study will assess the effectiveness, costs, and cost-effectiveness of 4 promising strategies to connect more primary care patients who smoke with evidence-based treatment to help them quit smoking. Results will be used to select an optimized package of interventions that seems to work especially well. The results of this research have the potential to suggest effective and efficient ways to reduce smoking prevalence by connecting more primary care patients who smoke to evidence-based care.

ELIGIBILITY:
Inclusion criteria:

* Primary care patient who receives care at one of the host family medicine or internal medicine clinics
* >17 years old
* Report smoking 7 of the last 7 days at enrollment
* Report smoking at least five cigarettes per day for at least 6 months at enrollment
* Able to speak and read English

Exclusion criteria:

* Opted out of Care Manager outreach at the most recent clinic visit or by phone
* Willing to quit smoking within 30 days (these patients will be referred for immediate treatment rather than enrolled in this study)
* Inability to use both C-NRT and varenicline due to a contraindication to both treatments at enrollment (allergic reactions, severe renal disease)
* Current treatment for schizophrenia or a psychotic disorder at enrollment
* History of suicide attempt in the past 10 years at enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Fiore, MD,MPH,MBA, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Center for Tobacco Research and Intervention, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available by UW-CTRI in accord with NCI data sharing policies.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after publication of primary outcome paper
Access Criteria: Prior written request to the PI.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 229 participants provided informed consent. A total of 210 consented participants completed the baseline assessments and randomization procedures and were considered fully enrolled in the trial.
Period: Overall Study
Arm/Group | Incentive,Tailored,Care Manage,Intensive Treatment | Incentive,Tailored,Care Manage,Standard Treatment | Incentive,Tailored,No Care Manage,Intensive Treatment | Incentive,Tailored,No Care Manage,Standard Treatment | Incentive,Untailored,Care Manage,Intensive Treatment | Incentive,Untailored,Care Manage,Standard Treatment | Incentive,Untailored,No Care Manage,Intensive Treatment | Incentive,Untailored,No Care Manage,Standard Treatment | No Incentive,Tailored,Care Manage,Intensive Treatment | No Incentive,Tailored,Care Manage,Standard Treatment | No Incentive,Tailored,No Care Manage,Intensive Treatment | No Incentive,Tailored,No Care Manage,Standard Treatment | No Incentive,Untailored,Care Manage,Intensive Treatment | No Incentive,Untailored,Care Manage,Standard Treatment | No Incentive,Untailored,No Care Manage,IntensiveTreatment | No Incentive,Untailored,No Care Manage,Standard Treatment
Started | 9 | 16 | 12 | 14 | 10 | 11 | 10 | 18 | 11 | 16 | 11 | 17 | 12 | 15 | 11 | 17
Completed | 5 | 15 | 12 | 13 | 9 | 11 | 10 | 16 | 11 | 16 | 10 | 15 | 9 | 13 | 10 | 16
Not Completed | 4 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 3 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1
Not completed — Death | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by PI | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Incentive,Tailored,Care Manage,Intensive Treatment | Incentive,Tailored,Care Manage,Standard Treatment | Incentive,Tailored,No Care Manage,Intensive Treatment | Incentive,Tailored,No Care Manage,Standard Treatment | Incentive,Untailored,Care Manage,Intensive Treatment | Incentive,Untailored,Care Manage,Standard Treatment | Incentive,Untailored,No Care Manage,Intensive Treatment | Incentive,Untailored,No Care Manage,Standard Treatment | No Incentive,Tailored,Care Manage,Intensive Treatment | No Incentive,Tailored,Care Manage,Standard Treatment | No Incentive,Tailored,No Care Manage,Intensive Treatment | No Incentive,Tailored,No Care Manage,Standard Treatment | No Incentive,Untailored,Care Manage,Intensive Treatment | No Incentive,Untailored,Care Manage,Standard Treatment | No Incentive,Untailored,No Care Manage,IntensiveTreatment | No Incentive,Untailored,No Care Manage,Standard Treatment | Total
Number analyzed (Participants) | 9 | 16 | 12 | 14 | 10 | 11 | 10 | 18 | 11 | 16 | 11 | 17 | 12 | 15 | 11 | 17 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.11 (13.20) | 53.81 (12.14) | 47.33 (13.42) | 48.57 (13.92) | 59.30 (14.16) | 47.46 (14.08) | 49.60 (12.80) | 49.67 (13.39) | 53.27 (11.23) | 48.88 (14.25) | 54.82 (12.15) | 48.18 (14.63) | 49.75 (14.25) | 47.73 (13.68) | 54.73 (12.41) | 52.12 (17.39) | 50.91 (13.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 8 | 11 | 8 | 8 | 7 | 11 | 7 | 10 | 9 | 12 | 9 | 9 | 11 | 9 | 147
  Male | 2 | 5 | 4 | 3 | 2 | 3 | 3 | 7 | 4 | 6 | 2 | 5 | 3 | 6 | 0 | 8 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 9 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 2 | 3 | 23
  Not Hispanic or Latino | 9 | 16 | 11 | 12 | 1 | 10 | 8 | 18 | 10 | 14 | 10 | 16 | 12 | 15 | 9 | 14 | 185
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 7 | 2 | 4 | 3 | 3 | 3 | 10 | 6 | 8 | 2 | 3 | 3 | 6 | 4 | 4 | 72
  White | 5 | 8 | 8 | 8 | 7 | 5 | 5 | 8 | 4 | 6 | 7 | 8 | 8 | 9 | 6 | 8 | 110
  More than one race | 0 | 1 | 1 | 1 | 0 | 2 | 2 | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 1 | 2 | 16
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 9 | 16 | 12 | 14 | 10 | 11 | 10 | 18 | 11 | 16 | 11 | 17 | 12 | 15 | 11 | 17 | 210

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Initiate Treatment Over 1 Year of Study Enrollment
Description: The operational definition of treatment initiation is completing at least 1 session of psychosocial treatment in an available smoking cessation treatment. The primary coding of this outcome will be binary (1=any treatment initiation, as defined above, over 1-year of study enrollment period, vs. 0=no evidence of treatment initiation).
Time Frame: 1 year
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Incentive,Tailored,Care Manage,Intensive Treatment | Incentive,Tailored,Care Manage,Standard Treatment | Incentive,Tailored,No Care Manage,Intensive Treatment | Incentive,Tailored,No Care Manage,Standard Treatment | Incentive,Untailored,Care Manage,Intensive Treatment | Incentive,Untailored,Care Manage,Standard Treatment | Incentive,Untailored,No Care Manage,Intensive Treatment | Incentive,Untailored,No Care Manage,Standard Treatment | No Incentive,Tailored,Care Manage,Intensive Treatment | No Incentive,Tailored,Care Manage,Standard Treatment | No Incentive,Tailored,No Care Manage,Intensive Treatment | No Incentive,Tailored,No Care Manage,Standard Treatment | No Incentive,Untailored,Care Manage,Intensive Treatment | No Incentive,Untailored,Care Manage,Standard Treatment | No Incentive,Untailored,No Care Manage,IntensiveTreatment | No Incentive,Untailored,No Care Manage,Standard Treatment
Number analyzed (Participants) | 9 | 16 | 12 | 14 | 10 | 11 | 10 | 18 | 11 | 16 | 11 | 17 | 12 | 15 | 11 | 17
Participants | 0 | 2 | 1 | 0 | 4 | 1 | 1 | 0 | 3 | 0 | 2 | 0 | 2 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Who Initiate Treatment Over 2 Years of Study Enrollment
Description: The operational definition of treatment initiation is completing at least 1 session of psychosocial treatment in an available smoking cessation treatment. The primary coding of this outcome will be binary (1=any treatment initiation, as defined above, over the 2-year study enrollment period, vs. 0=no evidence of treatment initiation).
Time Frame: 2 years
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Incentive,Tailored,Care Manage,Intensive Treatment | Incentive,Tailored,Care Manage,Standard Treatment | Incentive,Tailored,No Care Manage,Intensive Treatment | Incentive,Tailored,No Care Manage,Standard Treatment | Incentive,Untailored,Care Manage,Intensive Treatment | Incentive,Untailored,Care Manage,Standard Treatment | Incentive,Untailored,No Care Manage,Intensive Treatment | Incentive,Untailored,No Care Manage,Standard Treatment | No Incentive,Tailored,Care Manage,Intensive Treatment | No Incentive,Tailored,Care Manage,Standard Treatment | No Incentive,Tailored,No Care Manage,Intensive Treatment | No Incentive,Tailored,No Care Manage,Standard Treatment | No Incentive,Untailored,Care Manage,Intensive Treatment | No Incentive,Untailored,Care Manage,Standard Treatment | No Incentive,Untailored,No Care Manage,IntensiveTreatment | No Incentive,Untailored,No Care Manage,Standard Treatment
Number analyzed (Participants) | 9 | 16 | 12 | 14 | 10 | 11 | 10 | 18 | 11 | 16 | 11 | 17 | 12 | 15 | 11 | 17
Participants | 1 | 2 | 2 | 1 | 5 | 3 | 5 | 0 | 4 | 0 | 3 | 0 | 2 | 0 | 1 | 0

3. Secondary Outcome: Number of Participants Who Achieve Biochemically Verified Seven-day Point Prevalence Abstinence 2 Years Post-enrollment
Description: All study participants randomized to experimental condition will be asked to report on any smoking in the last 7 days at a follow-up phone interview 2 years after enrollment. Those claiming complete abstinence in the past 7 days at this follow-up interview will be asked to provide a saliva sample for biochemical verification of abstinence via cotinine testing. Participants who report abstinence in the last 7 days at this visit but have a cotinine level >10ng/mL or who do not have provide a cotinine result will be considered to be smoking. Missing data will be coded as not abstinent in primary, intent-to-treat analyses.
Time Frame: 2 years from enrollment
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Incentive,Tailored,Care Manage,Intensive Treatment | Incentive,Tailored,Care Manage,Standard Treatment | Incentive,Tailored,No Care Manage,Intensive Treatment | Incentive,Tailored,No Care Manage,Standard Treatment | Incentive,Untailored,Care Manage,Intensive Treatment | Incentive,Untailored,Care Manage,Standard Treatment | Incentive,Untailored,No Care Manage,Intensive Treatment | Incentive,Untailored,No Care Manage,Standard Treatment | No Incentive,Tailored,Care Manage,Intensive Treatment | No Incentive,Tailored,Care Manage,Standard Treatment | No Incentive,Tailored,No Care Manage,Intensive Treatment | No Incentive,Tailored,No Care Manage,Standard Treatment | No Incentive,Untailored,Care Manage,Intensive Treatment | No Incentive,Untailored,Care Manage,Standard Treatment | No Incentive,Untailored,No Care Manage,IntensiveTreatment | No Incentive,Untailored,No Care Manage,Standard Treatment
Number analyzed (Participants) | 9 | 16 | 12 | 14 | 10 | 11 | 10 | 18 | 11 | 16 | 11 | 17 | 12 | 15 | 11 | 17
Participants | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 2

4. Other Pre Specified Outcome: First Year Intervention Costs From Healthcare and Societal Perspectives
Description: The costs of implementing each intervention in the first year (minus research-related costs) will be computed from healthcare utilization, service, medication, administrative, and patient-report data. This outcome will be used to determine first-year costs of implementing each intervention component and highly promising intervention packages.
Time Frame: 1 year
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Second Year Intervention Costs From Healthcare and Societal Perspectives
Description: The costs of maintaining implementation of each intervention (minus research-related costs) will be computed from healthcare utilization, service, medication, administrative, and patient-report data. This outcome will be used to determine the costs of maintaining implementation of each intervention component and highly promising intervention packages.
Time Frame: 2 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Number of Participants Who Complete Intensive Treatment
Description: This outcome will be coded with a binary indicator of whether or not participants randomly assigned to have access to intensive treatment with C-NRT or varenicline completed a full round of treatment at any point over 2 years. Completion is defined as completing three phone counseling sessions.
Time Frame: 2 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Number of Participants Who Report Short-term Abstinence Following Smoking Cessation Treatment Initiation
Description: Self-reported 7-day point prevalence abstinence will be determined from participants who attempt to quit at 3 telephone follow-ups during an assisted quit attempt. At all 3 time-points, 7-day point-prevalence abstinence will be coded as binary (1=abstinent, not even a puff, in the past 7 days, per self-report, or 0=any smoking in the past 7 days), with missing treated as smoking in primary, intent-to-treat analyses.
Time Frame: 3, 12, and 26 weeks post-target quit day
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events were assessed systematically at follow-up phone interviews 6, 12, 18, and 24 months after enrollment and 3, 12, and 26 weeks after any target quit dates set by participants who initiated treatment in the study.
Arm/Group | Incentive,Tailored,Care Manage,Intensive Treatment | Incentive,Tailored,Care Manage,Standard Treatment | Incentive,Tailored,No Care Manage,Intensive Treatment | Incentive,Tailored,No Care Manage,Standard Treatment | Incentive,Untailored,Care Manage,Intensive Treatment | Incentive,Untailored,Care Manage,Standard Treatment | Incentive,Untailored,No Care Manage,Intensive Treatment | Incentive,Untailored,No Care Manage,Standard Treatment | No Incentive,Tailored,Care Manage,Intensive Treatment | No Incentive,Tailored,Care Manage,Standard Treatment | No Incentive,Tailored,No Care Manage,Intensive Treatment | No Incentive,Tailored,No Care Manage,Standard Treatment | No Incentive,Untailored,Care Manage,Intensive Treatment | No Incentive,Untailored,Care Manage,Standard Treatment | No Incentive,Untailored,No Care Manage,IntensiveTreatment | No Incentive,Untailored,No Care Manage,Standard Treatment
All-Cause Mortality (participants affected / at risk) | 1/9 | 1/16 | 0/12 | 0/14 | 0/10 | 0/11 | 0/10 | 0/18 | 0/11 | 0/16 | 0/11 | 2/17 | 0/12 | 1/15 | 0/11 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/9 | 5/16 | 1/12 | 1/14 | 3/10 | 3/11 | 2/10 | 6/18 | 3/11 | 2/16 | 3/11 | 5/17 | 3/12 | 9/15 | 4/11 | 3/17
Other Adverse Events (participants affected / at risk) | 1/9 | 0/16 | 1/12 | 1/14 | 1/10 | 1/11 | 1/10 | 0/18 | 1/11 | 0/16 | 1/11 | 0/17 | 1/12 | 1/15 | 1/11 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Incentive,Tailored,Care Manage,Intensive Treatment (N=9) | Incentive,Tailored,Care Manage,Standard Treatment (N=16) | Incentive,Tailored,No Care Manage,Intensive Treatment (N=12) | Incentive,Tailored,No Care Manage,Standard Treatment (N=14) | Incentive,Untailored,Care Manage,Intensive Treatment (N=10) | Incentive,Untailored,Care Manage,Standard Treatment (N=11) | Incentive,Untailored,No Care Manage,Intensive Treatment (N=10) | Incentive,Untailored,No Care Manage,Standard Treatment (N=18) | No Incentive,Tailored,Care Manage,Intensive Treatment (N=11) | No Incentive,Tailored,Care Manage,Standard Treatment (N=16) | No Incentive,Tailored,No Care Manage,Intensive Treatment (N=11) | No Incentive,Tailored,No Care Manage,Standard Treatment (N=17) | No Incentive,Untailored,Care Manage,Intensive Treatment (N=12) | No Incentive,Untailored,Care Manage,Standard Treatment (N=15) | No Incentive,Untailored,No Care Manage,IntensiveTreatment (N=11) | No Incentive,Untailored,No Care Manage,Standard Treatment (N=17)
Cardiac event or disease requiring hospitalization (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Including congestive heart failure, atrial fibrillation, myocardial infarction
Nervous system disorder requiring hospitalization or emergency care (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) — Including seizures
Surgery with hospitalization (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) — vascular, joint replacement
Respiratory illness requiring hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 1 (1) — Chronic obstructive pulmonary disease, asthma, and/or respiratory infections
Constipation, bowel obstruction, diarrhea requiring hospitalization (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Psychiatric hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pregnancy-related problems requiring hospitalization (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal or urinary issues (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hospitalization for gallstones (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
New cancer diagnoses (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscoskeletal injury prompting emergency care or hospitalization (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Endocrine-related hospitalization (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Unknown or other cause of death or hospitalization (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Incentive,Tailored,Care Manage,Intensive Treatment (N=9) | Incentive,Tailored,Care Manage,Standard Treatment (N=16) | Incentive,Tailored,No Care Manage,Intensive Treatment (N=12) | Incentive,Tailored,No Care Manage,Standard Treatment (N=14) | Incentive,Untailored,Care Manage,Intensive Treatment (N=10) | Incentive,Untailored,Care Manage,Standard Treatment (N=11) | Incentive,Untailored,No Care Manage,Intensive Treatment (N=10) | Incentive,Untailored,No Care Manage,Standard Treatment (N=18) | No Incentive,Tailored,Care Manage,Intensive Treatment (N=11) | No Incentive,Tailored,Care Manage,Standard Treatment (N=16) | No Incentive,Tailored,No Care Manage,Intensive Treatment (N=11) | No Incentive,Tailored,No Care Manage,Standard Treatment (N=17) | No Incentive,Untailored,Care Manage,Intensive Treatment (N=12) | No Incentive,Untailored,Care Manage,Standard Treatment (N=15) | No Incentive,Untailored,No Care Manage,IntensiveTreatment (N=11) | No Incentive,Untailored,No Care Manage,Standard Treatment (N=17)
Nausea or vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness or weakness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gas, constipation, or indigestion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Insomnia or vivid dreams (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest tightness or difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Changes in mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The target sample size to provide sufficient statistical power to detect hypothesized effects was N=1664. The trial was closed to recruitment after randomizing 210 participants because the recruitment model was not working as intended. We converted this trial into a pilot study and launched a new study that used clinic-level random assignment to evaluate different strategies to promote the reach of evidence-based tobacco treatment among adult primary care patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT04199117/Prot_SAP_001.pdf
  • Informed Consent Form (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT04199117/ICF_000.pdf